CLINICAL TRIAL: NCT07336979
Title: A Single-Arm, Phase Ⅱ Exploratory Study of Neoadjuvant Therapy With Paclitaxel Polymersomes for Injection Combined With Carboplatin and Adebelimab in the Treatment of Resectable Mucosal Melanoma
Brief Title: Paclitaxel Polymersomes + Carboplatin + Adebelimab: Neoadjuvant Phase Ⅱ Single-Arm Study for Resectable Mucosal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, xizhi wen, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-799-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Resectable Mucosal Melanoma
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel Polymersomes Combined with Carboplatin and Adebelimab (Experimental)
  Interventions: Drug: Paclitaxel Polymersomes Combined with Carboplatin and Adebelimab; Procedure: Radical Surgery

INTERVENTIONS:
Drug: Paclitaxel Polymersomes Combined with Carboplatin and Adebelimab — Chemotherapeutic agents are administered on Day 1 of each cycle: paclitaxel polymersomes for injection is given first, followed by carboplatin.Adebelimab injection is administered on Day 2 of each cycle.Patients will receive a maximum of 3 cycles of neoadjuvant chemotherapy combined with immunotherapy before surgery.Patients who are evaluated as resectable 3 weeks after the last cycle of chemotherapy will undergo radical surgery.
Procedure: Radical Surgery — Chemotherapeutic agents are administered on Day 1 of each cycle: paclitaxel polymersomes for injection is given first, followed by carboplatin.Adebelimab injection is administered on Day 2 of each cycle.Patients will receive a maximum of 3 cycles of neoadjuvant chemotherapy combined with immunotherapy before surgery.Patients who are evaluated as resectable 3 weeks after the last cycle of chemotherapy will undergo radical surgery.

SUMMARY:
The primary objective of this study is to evaluate the pathological response rate of neoadjuvant therapy with paclitaxel polymersomes for injection combined with carboplatin and adebrelimab in patients with resectable mucosal melanoma.Subjects will receive the combination therapy of paclitaxel polymersomes for injection, carboplatin and adebrelimab prior to surgery, with a treatment cycle of 3 weeks and a total of 3 cycles.After completing 3 cycles of treatment, subjects will undergo curative surgery. Pathologists will evaluate the surgically resected specimens to determine the status of pathological response, and immunohistochemical assays will be performed to assess the intensity of immune activation within the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Histopathologically confirmed resectable mucosal melanoma.
3. Subjects must provide 5 formalin-fixed paraffin-embedded (FFPE) tissue sections collected before treatment, or be willing to undergo needle biopsy for pathological tissue acquisition to facilitate pathological assessment.
4. ECOG (Performance Status, PS) score of 0-1.
5. No prior treatment with immune checkpoint inhibitors such as anti-CTLA-4, anti-PD-1, or anti-PD-L1 monoclonal antibodies.
6. No prior treatment with taxane-based drugs.
7. Presence of measurable lesions (per RECIST 1.1 criteria).
8. No history of immunosuppressant use within 6 months prior to enrollment.
9. Hematological and biochemical test results meeting the following criteria:

   i. Neutrophil count ≥ 1,500 × 10⁹/L; ii. Platelet count ≥ 100 × 10⁹/L; iii. Hemoglobin > 9.0 g/dL; iv. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min; v. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 3 × ULN; vi. Total bilirubin ≤ 1.5 × ULN.
10. Women of childbearing potential must have a negative serum or urine pregnancy test and agree to use an appropriate contraceptive method (barrier contraception or oral contraceptives).

Exclusion Criteria:

1. Presence of distant metastatic lesions.
2. Active autoimmune disease. Note: Patients with vitiligo, type 1 diabetes mellitus, or Hashimoto's thyroiditis with hypothyroidism who only require hormone replacement therapy may be enrolled if there is no evidence of significant disease recurrence.
3. Need for systemic corticosteroid therapy (> 10 mg prednisolone [or equivalent]/daily) or other immunosuppressant use within 14 days after enrollment. Note: Inhaled or topical corticosteroids, or adrenal hormone replacement therapy (> 10 mg prednisolone [or equivalent]/daily) are acceptable for patients without obvious autoimmune diseases.
4. Concurrent diagnosis of other malignant tumors requiring anti-tumor treatment. Note: Patients may be considered for enrollment if the other malignant tumor has achieved complete remission for 2 years or more and no additional anti-tumor treatment is required during the study period.
5. Patients who are medically, psychologically, or physically unable to complete the study or understand the information provided in the patient brochure, as assessed by the investigator.
6. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, or other drugs targeting T-cell costimulatory or immune regulatory pathways.
7. Prior chemotherapy with taxane-based drugs.
8. Positive HIV test result or confirmed diagnosis of acquired immunodeficiency syndrome (AIDS).
9. Known hypersensitivity to the study drugs.
10. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | 8 weeks
  The proportion of patients with less than 50% residual tumor cells in the surgically resected pathological specimens, including those who achieved pathological complete response (pCR), major pathological response (MPCR) and partial pathological response (pPR).

SECONDARY OUTCOMES:
overall response rate | 8 weeks
  The proportion of patients who achieve complete response (CR) or partial response (PR) evaluated according to the RECIST 1.1 criteria based on imaging examinations.
Surgical Resection Rate | 8 weeks
  calculated as the number of patients who underwent scheduled surgical resection divided by the number of enrolled patients.
Acute and Chronic Toxicities and Adverse Reactions | 8 weeks
relapse-free survival | 8 weeks
Assessment of Immune Activation Intensity in the Tumor Microenvironment | 8 weeks
  defined as the magnitude of changes in the proportions of CXCL13, CD4, CD8, CD19, and FOXP3-positive cells and the structural alterations of tertiary lymphoid organs (TLOs) in the tumor microenvironment before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No